CLINICAL TRIAL: NCT00718887
Title: A Comparative Study of the Week 12 Antiviral Efficacy and Safety of Switching to Entecavir vs. Continuing Adefovir Treatment in Adults With Chronic Hepatitis B and Suboptimal Response to Adefovir
Brief Title: Suboptimal Responders to Adefovir Switching to Entecavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AI463-171
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entecavir, 0.5 mg QD (Experimental)
  Interventions: Drug: Entecavir
- Adefovir, 10 mg QD/Entecavir, 0.5 mg QD (Other): Control
  Interventions: Drug: Adefovir/Entecavir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 0.5 mg, once daily (QD), 52 weeks
  Other Names: Baraclude; BMS-200475
  Arms: Entecavir, 0.5 mg QD
Drug: Adefovir/Entecavir — Tablets, Oral, 10-mg adefovir QD for 12 weeks followed by 0.5-mg entecavir QD for a maximum of 52 weeks
  Other Names: Baraclude; BMS-200475
  Arms: Adefovir, 10 mg QD/Entecavir, 0.5 mg QD

SUMMARY:
Switching to Entecavir will result in superior antiviral efficacy as compared to continuing with Adefovir in patients with a suboptimal response to Adefovir

ELIGIBILITY:
Inclusion Criteria:

* Chronic infection with hepatitis B virus (HBV)(detectable hepatitis B surface antibody (HBsAg) at screening and at least 24 weeks prior to screening, or detectable HBsAg for <24 weeks and negative for immunoglobulin M core antibody)
* Documentation of hepatitis B e antigen (HBeAg) positive or negative status
* Naive to nucleoside/nucleotide analogues, with the exception of adefovir
* Suboptimal response to adefovir treatment
* No lamivudine/telbivudine, entecavir, or adefovir resistance-associated substitutions at screening
* Male or female gender, aged 16 years and older
* Compensated liver function
* Serum alanine aminotransferase level <10*upper limit of normal at screening

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Evidence of decompensated cirrhosis
* Coinfection with HIV, hepatitis C virus, or hepatitis D virus
* Recent history of pancreatitis (within 24 weeks prior to the first dose of study medication)
* Chronic renal insufficiency, defined as a creatinine clearance <50 mL/min
* Current abuse of illegal drugs or alcohol, sufficient in the investigator's opinion to prevent adequate compliance with study therapy or to increase the risk of hepatotoxicity or pancreatitis
* Other serious medical conditions that might preclude completion of this study or that require chronic administration of prohibited medications
* Serum creatinine level >1.5 mg/dL; hemoglobin level <10.0 g/dL; platelet count <70,000/mm^3; absolute neutrophil count <1500 cells/mm^3; serum alpha fetoprotein level >100 ng/mL
* Except adefovir, any prior therapy with nucleoside or nucleotide analogue antiviral agents with activity against hepatitis B (eg, lamivudine, entecavir), or any other experimental anti-HBV antiviral, or any China Traditional Medicine
* Therapy with interferon, thymosin alpha, or other immunostimulators within 24 weeks of randomization
* Required chronic administration of medications that cause immunosuppression, that are associated with a high risk of nephrotoxicity or hepatotoxicity, or that affect renal excretion.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- China (7):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guiyang, Guizhou
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Nanchang, Jiangxi
  - Local Institution, Changchun, Jilin
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Shanghai, Shanghai Municipality

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 228 participants were enrolled, of which 169 were randomized. A total of 166 participants received treatment.
Groups:
- Entecavir, 0.5 mg QD: Participants with a pervious suboptimal response to adefovir received entecavir, 0.5 mg once daily (QD), for a maximum of 52 weeks.
- Adefovir, 10 mg QD/Entecavir, 0.5 mg QD: Participants with a previous suboptimal response to adefovir received adefovir, 10 mg QD, for 12 weeks. At 12 weeks, participants were switched to entecavir, 0.5 mg QD, for a maximum of 40 weeks.
Period: Overall Study
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Started | 89 (Participants who received treatment.) | 77 (Participants who received treatment.)
Completed | 84 (Continued in study after 48 weeks) | 68
Not Completed | 5 | 9
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Not identified | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD | Total
Number analyzed (Participants) | 89 | 77 | 166
Age Continuous [Median (Full Range); unit: Years] | 32.6 [16.9 to 62.4] | 34.1 [18.9 to 63.1] | 33.4 [16.9 to 63.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 75 | 67 | 142
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 89 | 77 | 166
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Hepatitis B Virus (HBV) DNA Level <50 IU/mL at Week 12 by Polymerase Chain Reaction Testing
Description: HBV DNA Level <50 IU/mL=approximately 300 copies/mL.
Time Frame: At Week 12 from Day 1
Population: Participants who were randomized and received at least
  1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Entecavir, 0.5 mg QD: Participants with a previous suboptimal response to adefovir received entecavir, 0.5 mg once daily (QD) for a maximum of 52 weeks.
- Adefovir, 10 mg QD: Participants with a previous suboptimal response to adefovir received adefovir, 10 mg QD for 12 weeks. At 12 weeks, participants were switched to entecavir, 0.5 mg QD, for a maximum of 40 weeks.
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD
Number analyzed (Participants) | 89 | 77
Percentage of participants | 5.6 | 0.0

2. Secondary Outcome: Percentage of Participants Who Achieved an HBV DNA Level <50 IU/mL at Week 48 by Polymerase Chain Reaction Testing
Description: HBV=hepatitis B virus. HBV DNA Level <50 IU/mL=approximately 300 copies/mL.
Time Frame: At Week 48 from Day 1
Population: Participants who were randomized and received at least
  1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Entecavir, 0.5 mg QD: Participants with a previous suboptimal response to adefovir received entecavir, 0.5 mg once daily (QD), for a maximum of 52 weeks.
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Number analyzed (Participants) | 89 | 77
Percentage of participants | 31.5 | 28.6

3. Secondary Outcome: Mean log10 Reduction From Baseline in Serum HBV DNA Level by Polymerase Chain Reaction Testing
Description: HBV=hepatitis B virus
Time Frame: At Weeks 12 and 48 from Day 1
Population: Participants who were randomized and received at least
  1 dose of study drug. n=number of evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Number analyzed (Participants) | 89 | 77
log10 IU/mL
  Week 12 (n=88, 77) | -2.5 (1.2) | -0.2 (1.1)
  Week 48 (n=87, 71) | -3.3 (1.5) | -3.2 (1.3)

4. Secondary Outcome: Percentage of Participants Who Achieved Normalization of Alanine Aminotransferase (ALT)
Description: ULN=upper limit of normal. ALT normalization= ≤1*ULN, among participants with baseline ALT >1*ULN
Time Frame: At Weeks 12 and 48 from Day 1
Population: Participants who were randomized, who received at least 1 dose of study drug, and whose ALT values were >1*ULN at baseline. n=number of evaluable participants.
Measure: Number; unit: Percentage of participants
Groups:
- Adeforvi, 10 mg QD/Entecavir, 0.5 mg QD: Participants with a previous suboptimal response to adefovir received adefovir, 10 mg QD, for 12 weeks. At 12 weeks, participants were switched to entecavir, 0.5 mg QD, for a maximum of 40 weeks.
Arm/Group | Entecavir, 0.5 mg QD | Adeforvi, 10 mg QD/Entecavir, 0.5 mg QD
Number analyzed (Participants) | 89 | 77
Percentage of participants
  Week 12 (n=51, 36) | 31.4 | 22.2
  Week 48 (n=51, 36) | 60.8 | 47.2

5. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B e Antigen (HBeAg) and Hepatitis B e (HBe) Seroconversion
Time Frame: At Weeks 12 and 48 from Day 1
Population: Participants who were randomized, who received at least 1 dose of study drug, and who were HBeAg-positive at baseline. n=number of evaluable participants.
Measure: Number; unit: Percentage of participants
Groups:
- Adefovir, 10 mg QD/Entecavir, 10 mg QD: Participants with a previous suboptimal response to adefovir received adefovir, 10 mg QD, for 12 weeks. At 12 weeks, participants were switched to entecavir, 0.5 mg QD, for a maximum of 40 weeks.
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 10 mg QD
Number analyzed (Participants) | 89 | 77
Percentage of participants
  HBeAG loss Week 12 (n=79, 72) | 3.8 | 6.9
  HBeAG loss Week 48 (n=79, 72) | 7.6 | 6.9
  HBe seroconversion Week 12 (n=79, 72) | 2.5 | 1.45
  HBe seroconversion Week 48 (n=79, 72) | 3.8 | 2.8

6. Secondary Outcome: Number of Participants With Hepatitis B s Surface Antibody (HBsAG) Loss and HBsAG Seroconversion
Time Frame: At Weeks 12 and 48 from Day 1
Population: Participants who were randomized and received at least
  1 dose of study drug. n=number of evaluable participants.
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Number analyzed (Participants) | 89 | 77
Participants
  Week 12 HBsAg loss | 0 | 0
  Week 48 HBsAg loss | 0 | 0
  Week 12 HBsAg seroconversion | 0 | 0
  Week 48 HBsAg seroconversion | 0 | 0

7. Secondary Outcome: Number of Participants With Genotypic Resistance to Entecavir
Time Frame: At Week 48 from Day 1
Population: Participants who were randomized and received at least
  1 dose of study drug. n=number of evaluable participants.
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Number analyzed (Participants) | 89 | 77
Participants
  At baseline | 0 | 0
  Week 48 | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events, Treatment-related AEs, Serious Adverse Events (SAEs), Treatment-related SAEs, Death as Outcome, Discontinuations Due to AEs, and Abnormalities in Laboratory Test Results (LTR) Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=possibly, probably, or certainly related to and of unknown relationship to study drug.
Time Frame: Continually from Day 1 through Week 48, and through 24-week follow-up period
Population: Participants who were randomized and received at least
  1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Number analyzed (Participants) | 89 | 77
Participants
  All AEs | 16 | 7
  Treatment-related AEs | 0 | 0
  SAEs | 1 | 0
  Treatment-related SAEs | 0 | 0
  Death | 0 | 0
  AEs leading to discontinuation | 1 | 0
  Abnormalities in LTR leading to discontinuation | 0 | 0

9. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Abnormalities in Laboratory Test Results
Description: Hematology testing assessed levels of hemoglobin, white blood cells, platelets, neutrophils, international normalized ration, red blood cells, lymphocytes, and monocytes.
Time Frame: Day 1 through Week 48
Population: Participants who were randomized and received at least
  1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Adefovir, 10 mg QD: Participants with a previous suboptimal response to adefovir received adefovir, 10 mg QD, for 12 weeks. At 12 weeks, participants were switched to entecavir, 0.5 mg QD, for a maximum of 40 weeks.
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD
Number analyzed (Participants) | 89 | 77
Percentage of participants
  Alanine aminotransferase | 9 | 5.2
  Aspartate aminotransferase | 2.2 | 0
  Hyperkalemia | 0 | 1
  Hematology | 0 | 0

ADVERSE EVENTS:
Arm/Group | Entecavir, 0.5 mg QD | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD
Serious Adverse Events (participants affected / at risk) | 1/89 | 0/77
Other Adverse Events (participants affected / at risk) | 8/89 | 9/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir, 0.5 mg QD (N=89) | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD (N=77)
Drug hepatitis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir, 0.5 mg QD (N=89) | Adefovir, 10 mg QD/Entecavir, 0.5 mg QD (N=77)
Alanine aminotransferase increased (Investigations) | 8 | 9
Aspartate aminotransferase increased (Investigations) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.